CLINICAL TRIAL: NCT02066207
Title: Open-label, Randomized, Multiple-dose, Crossover Study to Evaluate the Pharmacokinetic Interaction Between Fenofibrate and Atorvastatin in Healthy Male Volunteers
Brief Title: CKD-337 Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146DDI13024
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2014-03

CONDITIONS: Dyslipidemia (Fredrickson Type Ⅱa); Dyslipidemia (Fredrickson Type Ⅱb)
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fenofibrate (Experimental): Subjects received Fenofibrate
  Interventions: Drug: Fenofibrate
- Atorvastatin (Experimental): Subjects received Atorvastatin
  Interventions: Drug: Atorvastatin
- Fenofibrate and Atorvastatin (Experimental): Subjects received Fenofibrate and Atorvastatin
  Interventions: Drug: Fenofibrate; Drug: Atorvastatin

INTERVENTIONS:
Drug: Fenofibrate
  Arms: Fenofibrate; Fenofibrate and Atorvastatin
Drug: Atorvastatin
  Arms: Atorvastatin; Fenofibrate and Atorvastatin

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction between atorvastatin and fenofibrate in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male volunteer between 19 and 55 years old.
* BMI between 18.5 and 27.
* Able to participate in the entire trial
* Signed the informed consent form prior to study participation.

Exclusion Criteria:

* Clinically significant digestive system, cardiovascular system, respiratory system, endocrine system, hepatic system, renal system
* sit SBP < 100mmHg or sit SBP ≥ 150mmHg or sit DBP < 70mmHg or sit DBP ≥ 100mmHg
* Have acute infection history within 14 days
* Have a allergic disease of need to treat
* Have hypersensitivity reactions history for IP or any specific drugs.
* AST, ALT or Total bilirubin > UNL * 1.5
* Estimated GFR < 60 ml/min
* Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* A heavy smoker (cigarette > 10 cigarettes per day)
* A heavy alcohol consumer (alcohol > 140g/week)
* A heavy grapefruit consumer (more than 1cup per a day)
* Have a history of drug abuse or showed a positive for urine drug test.
* Administrated IP within 60 days prior to screening
* Rhabdomyolysis include of having a history or family history of genetic muscle diseases
* Positive for HIV antibody, HBsAg, HCV antibody test
* Previously donate whole blood within 60 days or component blood within 30 days
* Subject takes ethical drug or herbal medicine within 30 days
* Clinically significant laboratory test result
* An impossible one who participates in clinical trial by investigator's decision including other reason

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2014-04-07 (Actual); Study Completion 2014-05-29 (Actual)

PRIMARY OUTCOMES:
AUCt, Cmax,ss of fenofibric acid and atorvastatin | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 h

SECONDARY OUTCOMES:
Tmax,ss, Cmin,ss, t1/2, CL/Fss, Vd/Fss, %swing, Cav, %fluctuation | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea